CLINICAL TRIAL: NCT02753387
Title: Effect of Oral Preparation on Bacterial Colonization of the Pharyngeal Mucosa in Surgery of Head and Neck Cancer
Acronym: ORAL-ISO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC15_8923_ORAL-ISO
Record Dates: First submitted 2016-04-13; First posted 2016-04-27 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Bacterial Infection
Keywords: mouthwash; head and neck cancer; chlorhexidine; pathogens germs
MeSH Terms: conditions — Bacterial Infections; Head and Neck Neoplasms | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHLORHEXIDINE (Experimental): Patients will receive 1 preoperative oral preparation and 1 peroperative oral preparation of chlorhexidine
  Interventions: Drug: Chlorhexidine
- NaCl 0.9 % (Placebo Comparator): Patients will receive 1 preoperative oral preparation and 1 peroperative oral preparation of NaCl 0.9%
  Interventions: Device: NaCl 0.9 %

INTERVENTIONS:
Drug: Chlorhexidine — 4 mouthwashes during 30 seconds with Eludril Perio 10 ml and 1 application after intubation with Eludril Perio
  Other Names: Eludril Perio
  Arms: CHLORHEXIDINE
Device: NaCl 0.9 % — 4 mouthwashes during 30 seconds with NaCl 0.9 % 10 ml and 1 application after intubation with NaCl 0.9 %
  Arms: NaCl 0.9 %

SUMMARY:
Surgical site infections are an important health indicator for hospitals and a significant medico-economic issue.

The aim of the study is to assess the impact of chlorhexidine mouthwash performed before surgery on the bacterial colonization of the pharyngeal mucosa.

DETAILED DESCRIPTION:
The main objective is to reduce the number of patients with significant pathogenic bacterial colonization for pharyngeal mucosa at the end of the surgery. Oral flora is the same as the pharyngeal flora, so this suggests that the action of the oral mouthwash may also act in pharyngeal mucosa by buccopharyngeal communication.

Patients will be randomized into two groups :

* preoperative oral preparation with sodium chloride (NaCl) 0.9% (control group)
* preoperative oral preparation with chlorhexidine (experimental group)

A quantitative and qualitative analysis will be performed from samples collected during the surgery : before mouthwash (T0), after mouthwash (T1), before intubation in the operating room (T2), after intubation (T3), before incision (T4) and just before the end of the intervention on the mucosal scar (T5)

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of cancer regardless of histological type
* Surgical treatment requiring mucosal effraction regardless of the surgical approach;
* Patient over 18 years old;
* Oral cancer, oropharyngeal cancer, hypopharyngeal cancer or laryngeal cancer;
* Written and informed patient consent

Exclusion Criteria:

* Concomitant Vascular Interventions;
* Interventional radiology;
* Needing of second surgery at a same location during the 30 postoperative days);
* Cancer of the paranasal sinus, nasal cavity, skull base, salivary glands, skin,
* Neck dissection without mucosal effraction
* Thyroid or parathyroid surgery
* Size tumor forbidden tumor surgery
* Allergy to any tested product;
* Concurrent infection the day before or day of surgery
* Protected adults (guardianship) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with pharyngeal mucosa colonization (>=10^2 Colony Forming Unit (CFU)/ml of pathogen germs of the oral flora) at the end of the surgery | The day of the surgery
  The percentage of patients with pharyngeal mucosa colonization will be determined from the sample collected on the mucosal scar just before the end of the surgery (T5)

SECONDARY OUTCOMES:
Number of patients with a significant rate of pathogen germs (>=10^2 CFU/ml) at T1 | The day of the surgery
  The number of patients with a significant rate of pathogen germs will be determined from the sample collected after mouthwash (T1)
Type of oral germs | The day of the surgery
  The type of germs will be determined for all the samples collected during the surgery (i.e. before mouthwash (T0), after mouthwash (T1), before intubation in the operating room (T2), after intubation (T3), before incision (T4) and just before the end of the intervention on the mucosal scar (T5))
Number of positive cultures of pathogen germs | The day of the surgery
  The number of positive cultures of pathogen germs will be determined for all the samples collected during the surgery (i.e. before mouthwash (T0), after mouthwash (T1), before intubation in the operating room (T2), after intubation (T3), before incision (T4) and just before the end of the intervention on the mucosal scar (T5))
Kinetics of the number of CFU/ml | The day of the surgery
  The kinetics of the number of CFU/ml will be determined from all the samples collected during the surgery (i.e. before mouthwash (T0), after mouthwash (T1), before intubation in the operating room (T2), after intubation (T3), before incision (T4) and just before the end of the intervention on the mucosal scar (T5))
Number of CFU/ml of pathogens germs | The day of the surgery
  The number of CFU/ml of pathogens germs will be determined for all the samples collected during the surgery (i.e. before mouthwash (T0), after mouthwash (T1), before intubation in the operating room (T2), after intubation (T3), before incision (T4) and just before the end of the intervention on the mucosal scar (T5))
Surgical site infections rate in the postoperative month (standard definition of the Centers for Disease Control and Prevention, Atlanta) | 30 days
Number of patients who processed correctly preoperative mouthwash | The day of the surgery
Change in the number of CFU/ml of pathogen germs before and after intubation (T2-T3) | The day of the surgery
  The change in the number of CFU/ml of pathogen germs will be assessed using the samples collected before (T2) and after intubation (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Franck JEGOUX, PH, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No